CLINICAL TRIAL: NCT02085603
Title: SarCaBon: A Randomised Phase II Trial of Saracatinib Versus Placebo for Cancer-induced Bone Pain
Acronym: SarCaBon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STH16404; 2013-002505-62 (EudraCT Number)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Cancer
Keywords: advanced solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saracatinib (Active Comparator): Saracatinib at a dose of 125mg orally will be administered daily for four weeks.
  Interventions: Drug: Saracatinib
- Placebo (Placebo Comparator): Placebo tablet to be orally administered daily for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saracatinib
  Arms: Saracatinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to assess whether a drug called Saracatinib is helpful in controlling bone pain from cancer. The investigators do not know if it will be, so half of the patients in the study will receive the drug and half will get placebo. Saracatinib is a drug that has been tried in patients with many different forms of cancer. It seems to have effects in bone and so the investigators hope that it will have an effect in those with cancer that has spread to the bones.

DETAILED DESCRIPTION:
Controlling cancer pain in cancer patients can be very difficult as not all cancers respond to radiotherapy or chemotherapy and sometimes the sideeffects of strong painkillers, like morphine, can limit the dose of drug that can be given. The investigators have some evidence that a molecule called Src is involved in the development of cancer-induced bone pain. This study will use a drug, saracatinib that targets Src and will see if giving it to patients can reduce pain from cancer in the bones. The investigators will compare saracatinib to a placebo over a 4 week period in an estimated 62 patients. The investigators will measure whether the pain that patients report is less with saracatinib than placebo. The investigators will also measure how many painkillers people are taking before and after saracatinib/placebo, if pain thresholds have changed, if pain-related symptoms and quality of life have been improved and if saracatinib has a direct effect on the rate at which cancer breaks down bone.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent and willing to follow the study protocol.
* Age ≥ 16 years.
* Cytologically or histologically confirmed solid tumours of known primary site or multiple myeloma with painful bone metastases and poor control of bone pain in spite of pain medication including opioids
* WHO performance status ≤ 2
* Baseline BPI-SF score for pain on average ≥ 4 and ≤ 9 on a 0-10 numerical scale recorded on at least two separate days using the BPI-SF
* Adequate baseline haematological, hepatic and renal function, defined as follows:

  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Haemoglobin >9.0 g/dL (can be after transfusion)
  * Platelet count ≥ 100 x 109/L
  * Bilirubin ≤ 1.5 x ULN
  * ALT or AST ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
  * Creatinine ≤ 1.5 x ULN
* Ability to take and absorb oral medications.
* Female patients of childbearing potential (i.e. pre-menopausal females, females who have been menopausal for < 1 year and not surgically sterilized) must provide a negative pregnancy test (serum) ≤ 7 days before study treatment begins and must agree to practice effective contraceptive measures (oral contraceptive pill, intrauterine device or diaphragm with spermicide) plus condoms during the study and for 30 days after last dose of saracatinib.
* Male patients with a partner of child-bearing potential (who is not using an acceptable highly effective method of contraception) or a pregnant partner must use effective contraceptive measures (see 8) plus condoms during the study and for 3 months after the last dose of saracatinib. Patients should abstain from sperm donation during the study and for 3 months after the last dose of saracatinib.

Exclusion Criteria:

* Life expectancy < 3 months.
* Previous or planned radiotherapy at site of pain.
* Unstable cardiac disease in last 3 months.
* History of interstitial lung disease (bilateral, diffuse parenchymal lung disease) in view of known saracatinib-related pneumonitis.
* Unable to discontinue any medication with known moderate or potent inhibitory effect on CYP3A4, or or is a substrate of CYP3A4.
* Concomitant cytotoxic chemotherapy unless established on maintenance treatment for > 6 weeks (not in a clinical trial).
* Unable to understand written or spoken English as the primary outcome is dependent on completion of the BPI-SF questionnaire.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-01-21 (Actual)

PRIMARY OUTCOMES:
Is pain score lower after 4 weeks on treatment? | 4 weeks
  The primary outcome will be whether the patient's self-reported pain score is significantly lower after 4 weeks on treatment with saracatinib than after placebo.

SECONDARY OUTCOMES:
Does analgesic drug usage decreases when patients take saracatinib? | 4 weeks
  To determine if analgesic drug usage decreases when patients take saracatinib.
Does pain increase after treatment | 4 weeks
  To determine if pain thresholds at symptomatic sites increase after treatment with saracatinib.
Does symptoms and quality of life improve after treatment? | 4 weeks
  To determine if pain-related symptoms and quality of life are improved by saracatinib using the BPI-SF, EORTC QLQ-C30, EORTC BM-22 and GAPR questionnaires.
Is bone turnover further reduced by saracatinib? | 4 weeks
  To determine whether bone turnover is further reduced by saracatinib in patients already taking bisphosphonates or denosumab.
Safety of treatment | 4 weeks
  To determine the safety of saracatinib in this population by documenting adverse events and compliance.

OTHER OUTCOMES:
To calculate sample size for future trials | 4 weeks
  To resolve practical issues for the conduct of a future phase III RCT, such as the magnitude of the effect and its variability across the sample population, recruitment and attrition rates; and to inform the sample size calculation for a definitive trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Andrews, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Sheffield, South Yorkshire, United Kingdom